CLINICAL TRIAL: NCT01105676
Title: Vascular Malformations and Abnormalities of Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Beth Drolet, Professor and Vice Chairman of Pediatric Dermatology, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHW 08/204, GC 821
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Abnormality
Keywords: vascular malformation; vascular anomalies; abnormalities of growth; overgrowth; subjects with vascular malformations abnormalities of growth.
MeSH Terms: conditions — Congenital Abnormalities; Vascular Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single group single arm study (Experimental): Open no masking is used. All involved know the identity of the intervention assignment
  Interventions: Procedure: skin biopsy

INTERVENTIONS:
Procedure: skin biopsy — Two skin biopsies will be taken one time

SUMMARY:
To take part in this study you/your child have a vascular malformation, a type of blood vessel disorder whose cause is unknown.

The investigators will do this by looking at changes in the genes and proteins in the cells of the malformation as well as normal cells.

The investigators are doing this research because currently there is no known cause of vascular malformations and no way to know whether or not other health problems will occur in addition to the malformation. Through this research we hope to create standard methods for doctors to examine and treat people with vascular anomalies.

DETAILED DESCRIPTION:
If you/your child agree to participate

1. Informed consent and permission to use or disclose you/your child's health information for reserve purposes will be obtained by the research team. You will receive a copy of the consent form.
2. You/your child will be examined by a physician from the research team and interviewed about your medical background and condition every year for five years.
3. You/your child will have photographs taken of the affected area at each visit.
4. You/your child will have two, one time biopsies or skin samples taken by a dermatologist. Skin areas will be numbed with lidocaine and a 4 or 5 millimeter (or approximately 0.15 to 0.19 inch) sample will be taken in two different locations. The dermatologist taking the skin sample will use every effort to choose an area that can be covered by clothing or kept out of sight to others. The doctor will either use gelfoam or one stitch/suture per biopsy to seal off the area, which helps with healing and preventing bleeding. If a stitch is placed in the biopsy site, another visit about 7-10 days following the procedure will be necessary to remove the stitch.

5. You may still participate in the study if you consent to having only one biopsy taken of your affected (lesion) skin and not one of your unaffected (normal) skin.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 1 year of age
* Diagnosis of vascular malformation
* Each patient's authorized legal guardian must understand the nature of the study and must provide written informed consent. Each patient must also give assent to study participation given they have the cognitive capacity to do so.

Exclusion Criteria:

* Patients less than 1 year of age
* Vascular malformations likely to result in poor wound healing or located in areas of the body prone to significant scarring
* Individuals with vascular malformations and previous diagnosis of disseminated intravascular coagulopathy

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percent of growth over time | 5 years

SECONDARY OUTCOMES:
Patient specific gene and protein expression levels that can distinguish affected from unaffected tissue in patients. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Duffy, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Childrens Hospital of Wisconsin, Milwaukee, Wisconsin, United States